CLINICAL TRIAL: NCT00202995
Title: A Multi-Center, Randomized, Single-Blind, Parallel Group Study to Compare the Efficacy, Tolerability and Safety, of Copaxone® to That of High Dose Interferon (Betaseron® or Rebif®) in the Treatment of Relapsing Multiple Sclerosis Patients
Brief Title: Randomized Study Designed to Look at Disease Progression Using 2 Currently FDA Approved Drugs for the Treatment of RRMS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment decreased sample size No unexpected safety issues.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, Vice President, North American IR&D and Head of Global Clinical Operations, Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9013
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate; Interferon beta-1b; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Glatiramer Acetate 20 mg s.c. daily
  Interventions: Drug: Glatiramer Acetate
- 2 (Active Comparator): Betaseron 250 ug every other day or Rebif 44 ug 3 times a week
  Interventions: Drug: Betaseron; Drug: Rebif

INTERVENTIONS:
Drug: Glatiramer Acetate — 20 mg s.c. daily
  Arms: 1
Drug: Betaseron — 250 mg every other day
  Arms: 2
Drug: Rebif — 44 ug 3 times a week
  Arms: 2

SUMMARY:
Randomized study designed to look at the difference in relapse rates between patients remaining on their current interferon medication and those switched to Copaxone®

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of clinically definite MS with a relapsing disease course as determined by the Poser criteria
2. Patients must be on high dose interferon therapy (Betaseron® 250 µg or Rebif® 44 µg) for at least 1 year prior to study entry
3. Patients must have experienced at least one documented relapse during the past year prior to screening. Pseudo-relapses must be ruled out. A gadolinium enhancing lesion is not required.
4. Patients must be ambulatory, with a Kurtzke EDSS score between 0-5 inclusive
5. Patients must be between the ages of 18 and 50 years inclusive
6. Women of childbearing potential must practice an acceptable method of birth control. Acceptable methods include oral contraceptive, contraceptive patch, long-acting injectable contraceptive, double-barrier method (condom or IUD with spermicide), or partner's vasectomy
7. Patients must be relapse-free and off corticosteroids (IV or oral) for at least 30 days prior to the screening visit
8. Patients must be relapse-free and off corticosteroids between the screening and baseline visits
9. Patients must be willing and able to give written informed consent

Exclusion Criteria:

1. Use of experimental or investigational drugs, and/or participation in an investigational drug study within 6 months prior to study entry
2. Previous treatment with glatiramer acetate (injectable)
3. Previous treatment with immunomodulators (except IFNβ), immunosuppressive agents, IVIG, or plasma exchange in the 6 months prior to screening; previous treatment with cladribine in the past 2 years
4. Previous total body irradiation or total lymphoid irradiation
5. Chronic corticosteroid (IV, IM, and/or PO) treatment (more than 30 consecutive days) in the 6 months prior to study entry
6. Pregnancy or breastfeeding
7. Life-threatening or other clinically significant disease
8. Any condition which the investigator feels may interfere with participation in the study, including alcohol and/or drug abuse
9. A known sensitivity to gadolinium (gadolinium acid)
10. A known history of sensitivity to mannitol
11. Inability to successfully undergo MRI scanning

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2004-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to compare the total number of confirmed relapses experienced by patients randomized to maintain treatment on high dose IFN therapy compared to those who were switched to Copaxone® treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Brooks, Study Director — Teva Neuroscience, Inc.